CLINICAL TRIAL: NCT02863835
Title: Evaluation of Electrical Impedance Tomography for the Diagnosis of Chronic Rejection in Lung Transplants Recipients
Acronym: CLAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16/LO/0198
Record Dates: First submitted 2016-05-04; First posted 2016-08-11 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Transplantation, Heart-Lung; Chronic Lung Allograft Dysfunction; Bronchiolitis Obliterans Syndrome
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention 1 (Experimental): A 1:1 randomisation will be performed to decide the order of the administration of salbutamol and CPAP. All participants will receive both interventions in a cross-over fashion. Salbutamol nebulisation will be given during 15 minutes using 5mg of salbutamol. Assessments on CPAP will be performed at 3 different level of pressure.
  Each participant will then have continuous assessment of the following whilst self venting:
  * Spirometry - FEV1, FVC, MVV
  * Muscle strength measurements: MIP, MEP, SNIP
  * Borg scale, mMRC, Visual Analogue Scale for breathlessness
  * Electrical impedance tomography
  * EMGpara
  * Transcutaneous measurement of CO2 and 02 level
  * End-tidal CO2 monitoring
  * Pneumotachography
  Interventions: Other: EIT; Other: Salbutamol nebulisation and with CPAP

INTERVENTIONS:
Other: EIT — All participants will have continuous monitoring of EIT whilst self venting
Other: Salbutamol nebulisation and with CPAP — All participants will have continuous monitoring - salbutamol nebulisation will be given during 15 minutes using 5mg of salbutamol. Assessments on CPAP will be performed at 3 different level of pressure during this time.

SUMMARY:
Electrical impedance tomography (EIT) is non-invasive and provides functional imaging of the lung and it could be a useful tool to diagnose chronic lung allograft dysfunction (CLAD) and specially Bronchiolitis Obliterans Syndrome (BOS). Hence, for this study, the investigators aim to show that EIT would provide an accurate diagnostic CLAD with an ability to to distinguish BOS from Restrictive Allograft Syndrome (RAS) and to stage BOS accurately when compared to FEV1 the current gold standard. The investigators are also aiming to provide physiological data in lung transplant recipients with chronic rejection.

DETAILED DESCRIPTION:
Lung transplantation is the only treatment option available for patients affected by end-stage lung diseases such as chronic obstructive pulmonary disease (COPD), cystic fibrosis or idiopathic pulmonary fibrosis, not responding to maximal medical therapy. Despite the advance in the surgical techniques, immunosuppression treatment and prevention of acute cellular rejection episodes as well as opportunistic infections, the long terms outcomes following lung transplant remain unsatisfactory. Chronic lung allograft dysfunction (CLAD) is the first cause of long term mortality in lung transplant recipients responsible of 5 years mortality post-surgery of 50%. CLAD can lead to chronic respiratory failure and can presents in two different phenotypes: Restrictive forms of CLAD were all lung volumes are decreased (commonly called RAS, Restrictive Allograft Syndrome) that has been recently associated with antibodies mediated rejection. A more common form of obstructive CLAD has been identified as the well-known and defined Bronchiolitis Obliterans Syndrome (BOS). In patients with BOS, the progressive obliteration and a narrowing of the distal airways result in breathlessness, airflow obstruction and air trapping.

Currently, Forced Expiratory Volume at 1 second (FEV1) measurement is the gold standard to assess BOS severity. This test is non invasive and easily performed at bedside. Thus, it only gives a broad idea of the regional consequences of BOS as may be influenced by large airway obstructions. Chest computed tomography (CT) gives more detailed imaging of the regional consequences of BOS but is time-consuming and expose patients to radiations. Others imaging techniques such as ventilation/perfusion scintigraphy have been studied but cannot be performed at bedside.

As to date there is no curative treatment for BOS, preventive treatments such as long term azithromycin, bronchodilators, inhaled steroids or plasmapheresis have to be started at early stage of the disease to improve outcomes for the recipients Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air by the ventilator. It allows the assessment of these differences, which previously required the use of invasive equipment to obtain. Information is gained by repeatedly injecting small alternating electric currents (usually 5 mA) at high frequency of 50 - 80 kHz through a system of skin electrodes (usually 16) applied circumferentially around the thorax in a single plane between the 4th and 6th intercostal space. While an adjacent pair of electrodes 'injects' the current ('adjacent drive configuration'), all the remaining adjacent passive electrode pairs measure the differences in electric potential. A resistivity (impedance) image is reconstructed from this data by a mathematical algorithm using a two dimensional model and a simplified shape to represent the thoracic cross-section.

The resulting image possesses a high temporal and functional resolution making it possible to monitor dynamic physiological phenomena (e.g. delay in regional inflation or recruitment) on a breath by breath basis. It is important to realize that the EIT images are based on image reconstruction techniques that require at least one measurement on a well-defined reference state. All quantitative data are related to this reference and can only indirectly quantify (relative) changes in local lung impedance (but not absolute).

EIT can be used in mechanically ventilated patients to assess recruitment and to optimise ventilator settings to reduce risk of iatrogenic ventilator associated lung injury. To date, EIT has never been used in lung transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral lung transplant recipient
* Time from lung transplantation > 6 months
* A chest CT scan (HRCT) performed as part of their standard care in the last 3 months
* A bronchoscopy with BAL and Biopsies performed as part of their standard care in the last 3 months
* For group with CLAD: a drop in lung function assessed on FEV1 or FVC
* For group without CLAD: an unchanged lung function

Exclusion Criteria:

* Pregnancy
* Body mass index > 40kg/m2
* Significant physical or psychiatric comorbidity that would prevent compliance with trial protocol
* Allergy to salbutamol
* Patient with intra-bronchial or intra-tracheal metallic stent
* Evidence of acute infection or acute cellular rejection.

In addition 10 healthy volunteers will be recruited

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of chronic lung allograft dysfunction in lung transplant recipients identified with EIT | 1 day
  Using EIT to diagnose chronic lung allograft dysfunction in lung transplant recipients
Restrictive and obstructive phenotypes in recipients of lung transplants. | 1 day
  Using EIT to distinguish between restrictive and obstructive different phenotypes in recipients of lung transplants

SECONDARY OUTCOMES:
Change in EIT results following administration of salbutamol and CPAP | 1 day
  Following administration of salbutamol whilst using CPAP taking EITresults to determine if there is a change in the lungs
Correlation EIT results and chest-CT results | 1 day
  Comparing Lung measurements taken during the EIT test with the CT results of the participants to ascertain if there is any correlation
Neural respiratory drive (EMGpara) of lung transplant recipients | 1 day
  Comparing lung measurements taken during the EIT test with those taken during neural respiratory drive during the intervention
Correlation between EIT and neural respiratory drive results with breathlessness | 1 day
  Comparing lung measurements taken during the EIT test with the Neural respiratory drive results taken and the participants breathlessness
Correlation of EIT results found in obstructive and restrictive allograft syndrome | 1 day
  Comparing the obstructive allograft syndrome EIT results to the restrictive allograft syndrome results.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No